CLINICAL TRIAL: NCT03393325
Title: A Multicenter Observational Pilot Study on the Use of Tadalafil Delivra Cream in the Treatment of Raynaud's Phenomenon and Pain Associated With Digital Ulcers
Brief Title: Tadalafil-Delivra and Raynaud's Phenomenon
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decision. The study is not anticipated to start
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Delivra, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TAD-Sc-0001
Record Dates: First submitted 2017-12-22; First posted 2018-01-08 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Raynaud Phenomenon
MeSH Terms: conditions — Raynaud Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation of treatment with Tadalafil-Delivra — Tadalafil 2% in a Delivra base (Transdermal Application)

SUMMARY:
A 4-8 week observational feasibility study of the use of the use of Tadalafil-Delivra in the treatment of Reynaud's Phenomena (RP).

DETAILED DESCRIPTION:
To determine if the feasibility of conducting a future RCT using the chosen outcome assessments in RP patients at 2 Rheumatology clinics.

Study Design:

Observation of patients prescribed Tadalafil-Delivra 2% (Tad-Del) for the treatment of RP with defined feasibility objectives and data collection through efficacy and safety assessments. Study objectives are:

* At least 70% recruitment of eligible participants.
* 100% data collection from at least 70% of all enrolled subjects.
* Estimate the standard deviation(s) of all outcome assessments.

Setting/Participants:

Patients prescribed Tad-Del will be screened for study enrollment at 2 participating rheumatology clinics by the local research team. Participants that meet all the eligibility criteria will be enrolled in the study as subjects. Subjects will self-administer the medication as prescribed and return to the clinic for follow-up. Data will be collected on outcome assessments at: baseline, 1 week and at 4 to 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults of both genders, Age 18 to 75 years.
2. Patients with a confirmed diagnosis of Raynaud's Phenomenon (RP).
3. Written informed consent.
4. The presence of 1 or more digital ulcers (DU), that is not related to calcinosis, anywhere on a finger that is symptomatic for RP- defined as a VAS pain score of ≥25mm of 100mm Or 1 -3 fingers that are symptomatic for RP under standard of care treatment (SoC). Symptomatic is defined as a VAS pain score of ≥ 25mm of 100mm.
5. Prescribed, but not currently being treated with Tad-Del.
6. Maintenance of a stable background of prescribed treatment for RP including vasodilators, orally administered PDE5i and pain medication. Changes to administration of this concomitant medication will be documented in the case report form (CRF).

Exclusion Criteria:

1. Unwilling and/or incapable of adhering to the study procedures and follow-up schedule.
2. Use of other prescribed topical treatment for RP, such as nitrates.
3. Active infection of the index ulcer
4. Calcinosis at the site of the index ulcer
5. Received Iloprost or other prostacyclin treatment in the last 4 months.
6. Unsuitable for study participation as determined by the clinical investigator.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who have been prescribed Tad-Delivra for the treatment of primary or secondary Raynaud's Phenomenon with or without an active digital ulcer.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
VAS-100 of DU & RP severity over the previous week assessed by patient & MD | 28 days [this assessment has a window of an additional 28 days (Day 56) to be completed]
  Visual Analogue Scale (VAS) of the severity of Digital Ulcers (DU) and Raynaud's Phenomenon (RP). The physician (MD) and patient will each independently make their own assessment on a linear 10 cm VAS scale by making a mark on the line with a pen anywhere from the left anchor "0" (indicating no disease at all) to the right anchor "10" (indicating the most severe imaginable). Both the MD and patient will complete an individual scale for RP and DU. The distance of the mark from the left anchor "0" will be recorded in mm, divided by 10 and reported as a value from 0 to 10. A total of 4 VAS scales will be completed.

SECONDARY OUTCOMES:
Change in RP and DU interference in daily activities as measured by VAS-100 in SHAQ. | 28 days [this assessment has a window of an additional 28 days (Day 56) to be completed]
  Visual Analogue Scales for Raynaud's Phenomenon and Digital Ulcer interference in daily activities as measured by the patient. Both assessments are part of the Scleroderma Health Assessment Questionnaire (SHAQ). The patient will make an assessment on the linear VAS scale for each by making a mark on the line with a pen anywhere from the left anchor "Does not limit activities" to the right anchor "Very Severe limitation". The distance of the mark from the left to the right anchor will be measured in mm, divided by 10 and reported as a value from 0 to 10. There are two scales: 1 for Raynaud's Phenomena and the other for Digital Ulcer.
changes in the use of concurrent RP therapy and pain medications in patients treated with Tad-Del. | 28 days [this assessment has a window of an additional 28 days (Day 56) to be completed]
  Concomitant medication use at the end of treatment (day 28-56) will be compared with concomitant medication use at baseline with respect to daily dose administered.
All adverse Event experienced by the patient during study participation (1st to last visit) will be recorded. | 28 days [this assessment has a window of an additional 28 days (Day 56) to be completed]
  Adverse events will be summarized and reported at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Pope, MD PhD, Principal Investigator — St. Joseph's Health Care, London, ON
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No